CLINICAL TRIAL: NCT00337259
Title: Phase II Study of Gemcitabine in Patients With Advanced Stage Marginal Zone B-cell Lymphoma
Brief Title: Gemcitabine for Marginal Zone Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual and response less than expected on interim analysis
Sponsor: Asan Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Cheolwon Suh, ASCT team, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2006-60
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-Hodgkin's Lymphoma; Marginal Zone Lymphoma
Keywords: marginal zone lymphoma; gemcitabine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine (Experimental): * histologically confirmed marginal zone lymphoma
  * gemcitabine 1,250 mg/m2 on days 1 and 8 of each cycle, repeated every 3 weeks and continued for 6 cycles, until disease progression, withdrawal due to toxicity, or withdrawal of consent.
  Interventions: Drug: gemcitabine

INTERVENTIONS:
Drug: gemcitabine — D1 and 8, Gemcitabine 1250mg/m2 + NS 100ml MIV over 30min, every 3 weeks

SUMMARY:
Marginal zone lymphoma, one of the indolent lymphoma, is believed to be incurable with chemotherapy. Thus the investigators need a novel agent for marginal zone lymphoma. Gemcitabine has been tried as one of salvage chemotherapy regimen and has been shown to have anti-lymphoma activity. To the investigators' knowledge, there has been no trial of gemcitabine for marginal zone lymphoma. Thus the investigators made a plan to investigate the role of gemcitabine in marginal zone lymphoma.

DETAILED DESCRIPTION:
We designed a multi-center phase II trial of gemcitabine for advanced stage marginal zone B-cell lymphoma. Marginal zone lymphoma needs novel agent to improve clinical course by chemotherapy. Recent trials with new agents for indolent lymphoma shows promising results. Gemcitabine is known to have activity to non-Hodgkin's lymphoma and has less adverse effects than other new agents. With this background gemcitabine will be tried as a single agent for advanced marginal zone lymphoma.

Gemcitabine will be administered with 1,250mg/sq.m on days 1 and 8 every 3 weeks. Response will be assessed by IWC criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed marginal zone B-cell lymphoma
* Performance status (ECOG) ≤3
* Age ≥ 18
* At least one or more bidimensionally measurable lesion(s):

  * 2 cm by conventional CT
  * 1 cm by spiral CT

    * skin lesion (photographs should be taken)
    * measurable lesion by physical examination
* Laboratory values:

  * Cr < 2.0 mg% or Ccr > 60 ml/min
  * Transaminase < 3 X upper normal value
  * Bilirubin < 2 mg%
  * ANC > 1500/ul, platelet > 75,000/ul
* Informed consent
* Ann Arbor stage III or IV

Exclusion Criteria:

* Any other malignancies within the past 5 years except skin basal cell ca or CIS of cervix
* Serious comorbid diseases
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
response rate | CR+PR with study therapy

SECONDARY OUTCOMES:
safety and tolerability of the treatment | toxicity due to stdy drug

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No